CLINICAL TRIAL: NCT03510637
Title: ANRS 12332 HepNile : Evaluation of "Real Life" Efficacy and Safety of Antiviral Treatments Including New Direct Antiviral Agents Among Patients Treated for Chronic Hepatitis C (CHC) in Three National Treatment Centres in Cairo
Brief Title: "Real Life" Evaluation of Efficacy and Safety of Direct Antiviral Agents (DAAs) for the Treatment of Hepatitis C Virus in Egypt
Acronym: HepNile
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: ANRS 12332
Record Dates: First submitted 2018-04-13; First posted 2018-04-27 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C, Genotype 4, DAAs, Real life evaluation
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample (15 mL):
  * at inclusion,
  * at the End of Treatment (EOT)
  * 12 weeks after the end of treatment (only for patients who do not achieve a SVR).
  Samples (serum, plasma, DNA) stored in a dedicated biobank
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose of the ANRS 12332 HepNile study cohort is to assess in "Real-Life" condition the efficacy and the safety profile of new Direct Acting Antivirals (DAAs) introduced in the Egyptian National Treatment Programme for the treatment of Chronic Hepatitis C (CHC).

DETAILED DESCRIPTION:
Clinical trials are performed under optimal conditions where patients are highly selected with no co-morbidity, clinical supervision is provided by the best specialists in the field, and strict protocols are used to enhance patients' compliance. Thus, results may not be generalizable to real-world clinical practice.

Observational studies are now gaining attention, showing with previous treatments (combined pegylated interferon and ribavirin) a wide range of results in terms of treatment effectiveness (SVR from 21% to 63% overall), whereas related pivotal clinical trials had estimated SVRs between 54% and 63% overall.

Egypt is the first low/middle-income country where a national treatment program has been established on a large scale, allowing an evaluation that might be useful to itself and other similar countries. A real life evaluation will be particularly relevant now that new anti-viral drugs, direct-acting antivirals, are being introduced in Egypt.

ANRS 12332 HepNile cohort study will allow "in real life condition" the study of:

* Efficacy (cure rate) and safety of new HCV regimens introduced in Egypt
* Emergence of resistance variants for patients with virological breakthrough
* Factors associated with treatment failure
* Drug-Drug interactions
* Adherence to the treatment regimens

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA positivity
* 18 years =< Age =< 70 years
* Patients >= 65 years should undergo cardiological assessment prior to therapy by ECG echocardiography and cardiological consultation
* Effective contraception (Women of childbearing potential should use an effective contraception; Male patients and their female partners must also practice effective contraception) both during treatment and for the 3-months post-therapy); no breast-feeding
* Signed informed consent and willingness to participate in the study

Exclusion Criteria:

* Child C cirrhotic patients
* Platelet count > 50000/mm3
* Hepatocellular Carcinoma (HCC), except 6 months after intervention aiming at cure with no evidence of activity by dynamic imaging (CT or MRI)
* Extra-hepatic malignancy except after two years of disease-free interval (in case of lymphomas and chronic lymphatic leukemia, treatment can be initiated immediately after remission)
* Pregnancy or inability to use effective contraception
* inadequately controlled diabetes mellitus (HbA1C>9%)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a Chronic Hepatitis C and with prior approval from the Ministry of Health to begin HCV therapy
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2018-01-22 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Sustained Virological Response 12 weeks after the end of treatment (SVR12) | Post-treatment Week 12 (Week 24 or Week 36)
  Efficacy of treatment given by the proportion of patients with an HCV RNA undetectable 12 weeks after the completion of treatment.

SECONDARY OUTCOMES:
Proportion of patients with adverse reactions/events leading to dosage reduction and/or treatment discontinuation | End of Treatment Week 12 or Week 24
  Safety and tolerance profiles given by the proportion of patients with adverse reactions/events leading to dosage reduction and/or treatment discontinuation.
Adherence to treatment strategy | Post-treatment Week 12 (Week 24 or Week 36)
  Adherence given by the proportion of patients who have completed the treatment scheduled (defined by a patient who received 80% of drugs doses for 80% of the expected duration of therapy)
Resistance-Associated Variants (RAVs) | Post-Treatment Week 12 (Week 24 or Week 36)
  Assess the occurence of viral resistance patterns in HCV genotype 4 patients

CONTACTS AND LOCATIONS:
Overall Officials: Yehia Mohamed El Sayed El Shazly, MD, Principal Investigator — Ain Shams University; Arnaud Fontanet, MD, PhD, Principal Investigator — Institut Pasteur
Locations (3):
- Egypt (3):
  - El Fatemia El Kahera Centre, Cairo
  - National Hepatology and Tropical Medicine Institute, Cairo
  - New Cairo Hospital, Cairo

REFERENCES:
- [Background] Esmat G, El Kassas M, Hassany M, Gamil ME, El Raziky M. How to optimize HCV therapy in genotype 4 patients. Liver Int. 2013 Feb;33 Suppl 1:41-5. doi: 10.1111/liv.12059. PMID 23286845
- [Background] Doss W, Shiha G, Hassany M, Soliman R, Fouad R, Khairy M, Samir W, Hammad R, Kersey K, Jiang D, Doehle B, Knox SJ, Massetto B, McHutchison JG, Esmat G. Sofosbuvir plus ribavirin for treating Egyptian patients with hepatitis C genotype 4. J Hepatol. 2015 Sep;63(3):581-5. doi: 10.1016/j.jhep.2015.04.023. Epub 2015 May 1. PMID 25937436
- [Background] Obach D, Yazdanpanah Y, Esmat G, Avihingsanon A, Dewedar S, Durier N, Attia A, Anwar WA, Cousien A, Tangkijvanich P, Eholie SP, Doss W, Mostafa A, Fontanet A, Mohamed MK, Deuffic-Burban S. How to optimize hepatitis C virus treatment impact on life years saved in resource-constrained countries. Hepatology. 2015 Jul;62(1):31-9. doi: 10.1002/hep.27691. Epub 2015 Feb 27. PMID 25581111
- See also: Plan of action for the Prevention , Care & Treatment of Viral Hepatitis, Egypt, 2014-2018 — http://www.emro.who.int/images/stories/Hepatitis_action_plan.pdf?ua=1